CLINICAL TRIAL: NCT07164651
Title: Prospective Application Study of Intelligent Accelerated Magnetic Resonance Imaging in Children With Abdominal Pain
Brief Title: Intelligent Accelerated MRI for Pediatric Abdominal Pain
Acronym: IA-MRI
Status: Active, not recruiting | Type: Observational
Sponsor: Yaqi Shen，MD，PhD (Other)
Collaborators: United Imaging Healthcare (Unknown)
Responsible Party: Sponsor-Investigator, Yaqi Shen，MD，PhD, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202410027; 82471969 (Other Grant/Funding Number: National Natural Science Foundation of China (NSFC))
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Abdominal Pain
Keywords: Pediatric abdominal pain; Intelligent accelerated MRI; Image quality; Diagnostic accuracy; Motion artifacts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Pediatric patients who were undergoing MRE examination for abdominal pain
  Interventions: Other: Accelerated MRI scanning

INTERVENTIONS:
Other: Accelerated MRI scanning — All patients underwent MRI scans of the abdominal and pelvic regions on the uMR 790 scanner at Tongji Hospital's Optical Valley Campus. The scanning protocol included multiplanar ACS T2WI sequences, TACS T2WI sequences, and conventional T2WI sequences.
  ACS T2WI sequence: Used for preliminary motion artifact correction. TACS T2WI sequence: Employed for advanced motion artifact correction and provided dynamic images of organ movement.
  Conventional T2WI sequence: Served as the standard reference for comparison.

SUMMARY:
The goal of this observational study is to evaluate the effectiveness of an intelligent accelerated MRI technique in children with abdominal pain. The main question it aims to answer is:

Does the intelligent accelerated MRI reduce scan time while maintaining diagnostic accuracy in pediatric patients?

Participants will:

Receive an abdominal MRI scan using the accelerated protocol as part of their clinical evaluation.

Have their scan duration and image quality compared to conventional MRI standards.

DETAILED DESCRIPTION:
The goal of this prospective observational study is to evaluate the effectiveness and feasibility of an intelligent accelerated MRI scanning technique in pediatric patients presenting with abdominal pain. The main questions it aims to answer are:

Can the intelligent accelerated MRI technique achieve comparable or superior image quality to conventional MRI while significantly reducing scan time?

Does the accelerated scanning protocol reduce motion artifacts and improve diagnostic accuracy in pediatric patients?

Participants will:

Undergo an intelligent accelerated MRI scan of the abdomen as part of their diagnostic workup.

Have their scan duration, image quality, and diagnostic outcomes compared to historical or conventional MRI data (if available).

Why this study? Abdominal pain is a common pediatric complaint with diverse causes. While MRI is a non-invasive, radiation-free diagnostic tool, its utility in children is limited by long scan times and motion artifacts. This study investigates a novel intelligent accelerated MRI sequence that promises faster scans without compromising quality. Validating this technology in children could transform MRI's role in diagnosing abdominal pain by improving patient comfort, reducing sedation needs, and enhancing diagnostic accuracy.

Ethical approval: Conducted at Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, with oversight by the Institutional Ethics Committee.

Key innovation: Leveraging cutting-edge AI-driven acceleration to address pediatric imaging challenges. If successful, this approach could set a new standard for rapid, child-friendly MRI diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-18 years presenting with abdominal pain who have undergone abdominal CT examination.
* Children whose guardians voluntarily agree to MRI examination and sign written informed consent.

Exclusion Criteria:

* Children with contraindications to MRI (e.g., metal implants, severe claustrophobia) or those unable to cooperate with the examination.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consists of pediatric patients aged 3-18 years presenting with abdominal pain who have undergone a prior abdominal CT examination as part of their clinical evaluation. Eligible participants must have guardians who voluntarily consent to an additional MRI scan and provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Scan Time Reduction with Intelligent Accelerated MRI | During MRI scan procedure (single time point).
  Comparison of total scan time (minutes) for abdominal/pelvic MRI using the intelligent accelerated protocol (ACS-T2WI and TACS-T2WI sequences) versus conventional T2WI sequences, while maintaining diagnostic image quality (assessed by radiologists using a 5-point Likert scale).

SECONDARY OUTCOMES:
Diagnostic Accuracy of Accelerated MRI | Within 24 hours post-scan.
  Diagnostic concordance rate (%) between intelligent accelerated MRI and conventional MRI for identifying causes of abdominal pain (e.g., appendicitis, bowel obstruction), validated against final clinical/histopathological diagnoses.
Motion Artifact Reduction | During MRI scan procedure (single time point).
  Quantitative evaluation of motion artifacts in accelerated MRI scans (ACS-T2WI and TACS-T2WI) compared to conventional T2WI, scored by two blinded radiologists using a 4-point scale (1 = severe artifacts; 4 = minimal/no artifacts).

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Liu H, Deng D, Zeng W, Huang Y, Zheng C, Li X, Li H, Xie C, He H, Xu G. AI-assisted compressed sensing and parallel imaging sequences for MRI of patients with nasopharyngeal carcinoma: comparison of their capabilities in terms of examination time and image quality. Eur Radiol. 2023 Nov;33(11):7686-7696. doi: 10.1007/s00330-023-09742-6. Epub 2023 May 23. PMID 37219618
- [Result] Sui H, Gong Y, Liu L, Lv Z, Zhang Y, Dai Y, Mo Z. Comparison of Artificial Intelligence-Assisted Compressed Sensing (ACS) and Routine Two-Dimensional Sequences on Lumbar Spine Imaging. J Pain Res. 2023 Jan 28;16:257-267. doi: 10.2147/JPR.S388219. eCollection 2023. PMID 36744117
- [Result] Ni M, He M, Yang Y, Wen X, Zhao Y, Gao L, Yan R, Xu J, Zhang Y, Chen W, Jiang C, Li Y, Zhao Q, Wu P, Li C, Qu J, Yuan H. Application research of AI-assisted compressed sensing technology in MRI scanning of the knee joint: 3D-MRI perspective. Eur Radiol. 2024 May;34(5):3046-3058. doi: 10.1007/s00330-023-10368-x. Epub 2023 Nov 7. PMID 37932390
- [Result] Wang Q, Zhao W, Xing X, Wang Y, Xin P, Chen Y, Zhu Y, Xu J, Zhao Q, Yuan H, Lang N. Feasibility of AI-assisted compressed sensing protocols in knee MR imaging: a prospective multi-reader study. Eur Radiol. 2023 Dec;33(12):8585-8596. doi: 10.1007/s00330-023-09823-6. Epub 2023 Jun 29. PMID 37382615
- [Result] Wessling D, Herrmann J, Afat S, Nickel D, Almansour H, Keller G, Othman AE, Brendlin AS, Gassenmaier S. Application of a Deep Learning Algorithm for Combined Super-Resolution and Partial Fourier Reconstruction Including Time Reduction in T1-Weighted Precontrast and Postcontrast Gradient Echo Imaging of Abdominopelvic MR Imaging. Diagnostics (Basel). 2022 Sep 29;12(10):2370. doi: 10.3390/diagnostics12102370. PMID 36292057
- [Result] Chang PT, Yang E, Swenson DW, Lee EY. Pediatric Emergency Magnetic Resonance Imaging: Current Indications, Techniques, and Clinical Applications. Magn Reson Imaging Clin N Am. 2016 May;24(2):449-80. doi: 10.1016/j.mric.2015.11.009. Epub 2016 Feb 22. PMID 27150329
- [Result] Ata NA, Trout AT, Dillman JR, Tkach JA, Ayyala RS. Technical and Diagnostic Performance of Rapid MRI for Evaluation of Appendicitis in a Pediatric Emergency Department. Acad Radiol. 2024 Mar;31(3):1102-1110. doi: 10.1016/j.acra.2023.09.040. Epub 2023 Oct 19. PMID 37863782
- [Result] Sardar P, White CJ. Chronic mesenteric ischemia: Diagnosis and management. Prog Cardiovasc Dis. 2021 Mar-Apr;65:71-75. doi: 10.1016/j.pcad.2021.03.002. Epub 2021 Apr 24. PMID 33901516
- [Result] Gans SL, Pols MA, Stoker J, Boermeester MA; expert steering group. Guideline for the diagnostic pathway in patients with acute abdominal pain. Dig Surg. 2015;32(1):23-31. doi: 10.1159/000371583. Epub 2015 Jan 28. PMID 25659265
- [Result] Durgun Y, Yurumez Y, Guner NG, Aslan N, Durmus E, Kahraman Y. Abdominal Pain Management and Point-of-care Ultrasound in the Emergency Department: A Randomised, Prospective, Controlled Study. J Coll Physicians Surg Pak. 2022 Oct;32(10):1260-1265. doi: 10.29271/jcpsp.2022.10.1260. PMID 36205268
- [Result] Murphy LK, Suskind DL, Qu P, Zhou C, Gashi K, Kawamura JS, Palermo TM; ImproveCareNow Pediatric IBD Learning Health System, as stipulated by ICN. Abdominal Pain After Pediatric Inflammatory Bowel Disease Diagnosis: Results From the ImproveCareNow Network. J Pediatr Gastroenterol Nutr. 2020 Dec;71(6):749-754. doi: 10.1097/MPG.0000000000002933. PMID 32910089
- [Result] Smith J, Fox SM. Pediatric Abdominal Pain: An Emergency Medicine Perspective. Emerg Med Clin North Am. 2016 May;34(2):341-61. doi: 10.1016/j.emc.2015.12.010. PMID 27133248